#### Cover Letter:

All enclosed below documents are part of the clinical trial NCT03536819

Study Name: Radio-frequency rejuvenation for pelvic floor and vagina

Protocol No.: DO607404A

Document date: September 20, 2017

**SPONSOR**: InMode Ltd.

Tabor House

Industrial Park South

Yokneam 20692 ISRAEL

POB 44

Tel +972-4-9097309

Fax +972-4-9096310

**Study Title** 

Radio-frequency rejuvenation for pelvic floor and vagina

Protocol No

Sponsor

InMode MD Ltd.

Investigational Product

The Votiva system has been cleared by the United States Food and Drug Administration (FDA) for sexual dysfunction and pelvic floor relaxation.

Study Design

Prospective clinical study.

Study Objectives

#### Primary Objective:

Evaluate the effects of radiofrequency on pelvic floor strength as measured by intentional muscle contraction.

#### Secondary Objective:

- Evaluate the effects on subjective symptoms associated with pelvic floor weakness, including urinary symptoms, sexual function, sensitivity to climax, colorectal-anal symptoms
- -Evaluate patients' subjective efficacy and change of quality of life treatment.
- Evaluate patients' satisfaction at follow up visit

#### Primary Endpoints

- Completion of all proposed visits.
- Voluntary withdrawl of the patient at any time.

#### Efficacy Endpoints

Comparison of measurements and patient reporting via validated questionnaires after treatments to baseline, will quantify the effects of Forma V on pelvic floor laxity and the associated symptoms.

#### Objective measurements:

- -Genitalia(vaginal and labia) condition and intentional muscle contraction will be evaluated at baseline, before each treatment and at follow up visits (8 weeks after each treatment). Visits 2, 4 and 6.
- -Physical measurements of vagina, vulvar and perineal areas will be measured according to POP-Q guidelines. (Appendix 11.0) Visits 2, 4 and 6.

#### Subjective measurements:

 Subjective assessment of efficacy on sexual dysfunction symptoms, using the Female Sexual Function Index (FSFI) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) questionnaire (Appendix 6.0, 9.0) at visits 1, 5 and 7.

- Subjective assessment of efficacy on Urinary Incontinence symptoms
  using the International Consultation on Incontinence Questionnaire (ICIQ)
  and Questionnaire for Female Urinary Incontinence (QUID) (Appendix 7.0)
  at visits 1, 5 and 7.
- Subjective assessment of quality of life change using Pelvic Floor Impact Questionnaire (PFIQ-7) (Appendix 8.0) at visits 1, 5 and 7.
- Subjective assessment of improvement of pelvic organ prolapse, colorectal-anal disease or urinary distress as measured by the Pelvic Floor Distress Inventory Questionnaire (PFDI-20) (Appendix 10.0) at visits 1, 5, 7.

#### Safety Monitoring Procedures

- Observation, assessment and recording of reactions by the investigator.
- Evaluations will be done immediately after each treatment and at the followup visit. The frequency, severity and causality of all reactions will be recorded.
- Possible Votiva reactions are listed under potential risks.
- Severe and persistent reactions are reportable as adverse events.

# Patient Population and Sample Size

At least 20 female subjects ages 35-75 selected based on evaluation of symptoms including the following: urinary incontinence, pelvic floor laxity.

#### **Study Duration**

Study duration for each subject is approximately four months (including screening, 2 treatment sessions 8 weeks apart and a follow-up visit at 8 weeks post last treatment.

Overall study duration will be approximately 12 months, depending on the subject recruitment rate.

Each subject will undergo 7 study visits including screening, 2 treatment and 1 follow-up visit.

#### Visit 1: Midwest Plastic Surgery-Evaluation

- Screening will be performed to determine subject eligibility as well as to collect all of the required medical information and obtain signed Informed Consent.
- Baseline photographs of the treatment area will be taken
- Pre-procedure questionnaires will be completed at this time
- Time required 1.5 hours

#### Visit 2: Antares Institute-Evaluation

- A complete pelvic floor assessment will be performed including but not limited to the following: measurement of internal and external pelvic floor contraction, measurement of vaginal canal length and diameter, measurement of the introitus, and length of the labia majora and minora. Measurements will be obtained following POP-Q protocol
- This visit will confirm inclusion criteria based on measurements.
- Time required: 1.5hrs

#### **Visit 3:** Midwest Plastic Surgery – 1<sup>st</sup> treatment

- Internal and external FormaV treatment
- Photographs of the treatment area will be taken after the procedure.
- Time required: 45 minutes

#### Visit 4: Antares Institute Follow-up visit – 8 weeks following first treatment

- A complete pelvic floor assessment will be performed including but not limited to the following: measurement of internal and external pelvic floor contraction, measurement of vaginal canal length and diameter, measurement of the introitus, and length of the labia majora and minora. Measurements will be obtained following POP-Q protocol.
- Time required: 15 minutes

### **Visit 5:** Midwest Plastic Surgery – 2<sup>nd</sup> treatment

- Photographs of the treatment area will be taken before and after the procedure.
- Questionnaires will be completed.
- Time required: 45 minutes

### Visit 6: Antares Institute Follow-up visit – 8 weeks following second treatment

 A complete pelvic floor assessment will be performed including but not limited to the following: measurement of internal and external pelvic floor contraction, measurement of vaginal canal

length and diameter, measurement of the introitus, and length of the labia majora and minora. Measurements will be obtained following POP-Q protocol

- Time required: 15 minutes

Visit 7: Midwest Plastic Surgery – Follow-up visit – 8 weeks following second treatment

- Photographs of the treatment area will be taken
- Questionnaires will be completed
- Time required: 45 minutes
- After each treatment and at all visits, adverse events will be recorded. Duration of each treatment visit is specified.

### Main Eligibility Criteria

#### <u>Inclusion Criteria</u>

- Adult females between the ages of 35-75, seeking treatments for pelvic floor relaxation syndrome or atrophic vaginitis, which include but are not limited to: pelvic floor laxity, decreased muscle contraction in the pelvic floor, urinary incontinence, sexual dysfunction.
- Participants must have an evaluation by the Pelvic Floor Physical Therapists at Antares Institute. All participants must have a minimum of 30% below average reading on initial assessment of internal or external pelvic floor contraction in order to be included in the study.
- Negative PAP smear and pelvic exam done within last 1 year.
- The patients should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, (including the permission to use photography).
- The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other treatment methods in the treatment areas such surgeries, CO2 treatment, other radiofrequency treatments and fillers injections for the last 12 months and during the entire study period.
- Dr. Kouris will be available for consultation as needed throughout the course of the study. He will also review all documentation as needed.

#### Exclusion Criteria:

- Internal defibrillator, pacemaker, bladder stimulator or any other implanted electrical device anywhere in the body
- Permanent metal implant in the treatment area
- History of pelvic floor radiation
- Any surgery in the treatment area in the last 3 months
- Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
- Pregnancy and nursing

- Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
- Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, <u>may be treated only following a prophylactic</u> <u>regimen.</u>
- Poorly controlled endocrine disorders, such as diabetes, thyroid dysfunction, polycystic ovary and hormonal virilization
- Any active condition in the treatment area, such as but not limited to open sores, psoriasis, eczema, vitiligo, herpes and rash.
- History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin
- Severe concurrent conditions, such as cardiac disorders, sensory disturbances.
- Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
- Diseases that may be stimulated by light, such as epilepsy, lupus and urticaria.
- -Any other previous treatments in the vaginal or perineal area, such as CO2 laser or RF performed on the same area.
- -Any surgical procedure in the vaginal area within the past 12 months.
- -Recent tan from sun, sunbeds or chemicals or planned excessive sun exposure.
- -As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient

## Alternative therapies

-Participation in this study is not required to receive treatment for pelvic floor relaxation or sexual dysfunction. Patients may receive treatments without participating in the study. Patients may also utilize other methods of treatment including but not limited to Pelvic floor physical therapy, CO2 treatment, or other radiofrequency treatments.